CLINICAL TRIAL: NCT04192942
Title: Protocol of Management of Major Pediatric Burn in Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed elsayed tawfik, Official investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: major burn in childern
Record Dates: First submitted 2019-10-14; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Intensive Care Units

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intensive care management (Experimental): Administration of childern with major burn in intensive care to improve out comes
  Interventions: Other: protocol of management of major burn in intensive care unit

INTERVENTIONS:
Other: protocol of management of major burn in intensive care unit — primary assessment first aid management laboratory investigation radiological investigation surgical intervention

SUMMARY:
Decrease mortality and morbidity in major pediatric burns

DETAILED DESCRIPTION:
The goals of initial patient management include preservation of overall homeostasis while appreciating the physiologic challenges that the burn injury poses to the body. Major burn injury not only results in local damage from the inciting injury, but in many cases results in multisystem injury. Initial efforts are focused on resuscitation, maintaining hemodynamic stability, and airway management. Intermediate efforts are focused on managing the multi-organ failure that results from systemic inflammatory mediators that result in diffuse capillary leak and surgical therapy. Finally, efforts shift to issues with chronic wound healing, pain management, restoration of functional capabilities, and rehabilitation.. Burn injury in children continues to be a major epidemiologic problem around the globe. Nearly a fourth of all burn injuries occur in children under the age of 16, of whom the majority are under the age of five This provides a team of pediatricians, surgeons, anesthesiologists, intensivists, nurses, respiratory therapists, and other healthcare providers with a unique opportunity to make a multidisciplinary collaborative effort.

ELIGIBILITY:
Inclusion Criteria:

* age below 18 year
* children with burn between 20% to 50% of total body surface area
* recent burn within 48 hour

Exclusion Criteria:

* old burn over 48 hour after injury -burnt surface area less than 20% of total body surface area - -
* burnt surface area more than 50% of total body surface area
* old age over 18 year

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Changing mortality rate | baseline
  Change mortality rate to lowest degree which due too severe burn less than 20% of childern with major burn

SECONDARY OUTCOMES:
Changing hospital stay time | Baseline
  Hospital stay less than 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Azza Eltayeb, Professor, Study Director — Professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krishnamoorthy V, Ramaiah R, Bhananker SM. Pediatric burn injuries. Int J Crit Illn Inj Sci. 2012 Sep;2(3):128-34. doi: 10.4103/2229-5151.100889. PMID 23181206
- [Background] Williams FN, Herndon DN, Hawkins HK, Lee JO, Cox RA, Kulp GA, Finnerty CC, Chinkes DL, Jeschke MG. The leading causes of death after burn injury in a single pediatric burn center. Crit Care. 2009;13(6):R183. doi: 10.1186/cc8170. Epub 2009 Nov 17. PMID 19919684